CLINICAL TRIAL: NCT06971276
Title: Assessing the Utility of Plasma ctHPVDNA for Anal Cancer Screening
Acronym: SCAN-LITE
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Daniel L. Faden, MD, Assistant Professor, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 18-649
Record Dates: First submitted 2025-05-05; First posted 2025-05-14 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-05

CONDITIONS: Anal Dysplasia
Keywords: HPV; Liquid biopsy; Anal cancer; Anal intraepithelial neoplasia; Early cancer detection; HPV-DeepSeek; NGS
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, and tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Anal cancer: Screening patients diagnosed with anal squamous cell carcinoma (ASCC)
- AIN3: Screening patients diagnosed with anal intraepithelial neoplasia 3 (AIN3)
- AIN2: Screening patients diagnosed with anal intraepithelial neoplasia 2 (AIN2)
- AIN1: Screening patients diagnosed with anal intraepithelial neoplasia 1 (AIN1)
- HPV Infection: Screening patients diagnosed with HPV infection (no lesion)
- Controls: Screening patients diagnosed negative for HPV and control patients from the general population.

SUMMARY:
The study is to test a liquid biopsy assay for screening and classifying anal dysplasia from blood.

DETAILED DESCRIPTION:
Anal squamous cell carcinoma, despite being considered as a rare cancer, has seen a steady rise in incidence over the past three decades. Recent evidence from the Anal Cancer-HSIL Outcomes Research (ANCHOR) study demonstrated benefits of treating anal high-grade squamous intraepithelial lesion (HSIL), highlighting the importance of screening anal cancers and high-grade precancers. Current anal cancer screening starts with HPV testing and/or cytology for primary screening, followed by high-resolution anoscopy (HRA) with biopsy for confirmatory diagnosis. However, the poor specificity of HPV testing and the extremely limited capacity of HRA urges the development of new screening approaches for identifying anal high-grade precancers and cancers. Blood circulating tumor HPV DNA (ctHPVDNA) is an emerging non-invasive biomarker for screening and treatment monitoring of HPV-associated cancers, but its significance in anal cases remains underexplored. Here the investigators use an ultrasensitive HPV whole genome sequencing assay to test the hypothesis that anal precancers are detectable in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Past or current anal HPV-positive population undergone anal dysplasia screening.
* Control patients from the general population.

Exclusion Criteria:

* Not meeting inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergone screening for anal dysplasia and control patients from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Cancer Developmental Stage | Periprocedural
  Anal dysplasia screening results based on tissue biopsy collected at time of the visit or clinical diagnosis when biopsy is not available.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L. Faden, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Department of Infectious Diseases, Mass General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No